CLINICAL TRIAL: NCT00373009
Title: Prevention of Low Back Pain in the Military. A Randomized Clinical Trial
Brief Title: Prevention of Low Back Pain in the Military
Acronym: POLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PR054098
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: Low back pain; Primary prevention; Secondary prevention; Lumbar stabilization; Psychosocial education
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Core stabilization and psychosocial education (Experimental): A core stabilization exercise program (CSEP) is used in this group and has sound biomechanical and anatomical rationale. In addition, a psychosocial education program (PSEP) will be used for this group.
  Interventions: Behavioral: Core stabilization and psychosocial education
- Core stabilization exercise only (Active Comparator): A core stabilization exercise program (CSEP) is used in this group and has sound biomechanical and anatomical rationale.
  Interventions: Behavioral: Core stabilization exercise only
- Psychosocial education class only. (Active Comparator): A psychosocial education program (PSEP) will be used in this group.
  Interventions: Behavioral: Psychosocial education class only
- Traditional Army training (Other): Traditional Army training will be used in this group.
  Interventions: Behavioral: Traditional Army training

INTERVENTIONS:
Behavioral: Traditional Army training — As usual training for Soldiers
  Arms: Traditional Army training
Behavioral: Core stabilization exercise only — Core stabilization exercise
  Arms: Core stabilization exercise only
Behavioral: Psychosocial education class only — Psychosocial education class
  Arms: Psychosocial education class only.
Behavioral: Core stabilization and psychosocial education — Includes both core stabilization training and psychosocial education class
  Arms: Core stabilization and psychosocial education

SUMMARY:
We are studying whether specific back exercise and education programs effectively limit the development of chronic low back pain in Soldiers in the United States Army. These programs represent the current best evidence for prevention of low back pain from an exercise and education perspective. This innovative study will investigate whether a combination of evidence-based exercise and education programs effectively decreases the impact of chronic low back pain, when compared to individual evidence-based exercise and education programs, or a traditionally implemented exercise program.

DETAILED DESCRIPTION:
Background: Low back pain (LBP) is a musculoskeletal condition that accounts for significant pain and disability, and consumes substantial medical and occupational costs annually. Specific to the United States Armed Forces, LBP was the second most common reason to seek healthcare and affects over 150,000 active duty Soldiers annually (MSMR 2003). Soldiers in the U.S. Army with LBP have the highest risk of disability 5 years after their injury. Furthermore, a military review suggests that LBP was the most common condition bringing about a medical board, with lifetime direct compensation costs estimated to reach into the billions of dollars. Therefore, reduction of disability from LBP is a significant research priority for the military.

Reduction of disability from LBP has been divided into 2 separate phases - primary and secondary prevention. Primary prevention refers to interventions and strategies that are implemented before a low back injury occurs.8 Primary prevention reduces LBP related disability by reducing the total number of people who eventually experience an episode of LBP. Secondary prevention refers to interventions and strategies that are implemented during the acute episode of low back injury, before chronic symptoms occur.9 Secondary prevention reduces LBP related disability by reducing the number of people who eventually experience chronic disability from LBP. We are proposing an innovative approach to LBP prevention by combining primary and secondary prevention strategies that have the potential to limit the development of chronic LBP in Soldiers.

The primary prevention strategy is a core stabilization exercise program (CSEP). The CSEP used in this study has sound biomechanical and anatomical rationale, and has demonstrated its clinical efficacy by preventing future recurrence of LBP. However, this CSEP has not been previously investigated for primary prevention of LBP in healthy Soldiers. The secondary prevention strategy is a psychosocial education program (PSEP). The PSEP used in this study has sound theoretical rationale. It has also demonstrated its clinical efficacy by favorably altering LBP beliefs, as well as limiting the eventual severity of LBP episodes.

These programs (individually or in combination) have not been investigated for prevention of chronic LBP in healthy Soldiers. Therefore, we will train healthy Soldiers in the United States Army in CSEP, PSEP, or combined CSEP/PSEP. We will compare the preventative effects of these exercise and education programs to an already implemented traditional exercise program (TEP).

Objective/Hypothesis: The purpose of this study is to determine if a combined prevention program is more effective at limiting the development of chronic LBP when compared to the effects of individual evidence-based prevention programs, or a traditional exercise program

Specific Aims Specific Aim 1: We will determine if a combined prevention program consisting of CSEP and PSEP prevents the development of chronic LBP. During advanced individual training (AIT), United States Army Soldiers will be randomly assigned to receive 1 of 4 prevention programs. Soldiers will be followed monthly to measure LBP occurrence and severity during 2 years of active duty with a web-based data collection system managed at the University of Florida.

Specific Aim 2: We will determine if the CSEP results in favorable changes in specific core musculature associated with reducing LBP. The CSEP activates specific core musculature that are important in preventing LBP. We will use real-time ultrasound imaging to document changes in core musculature that occur during AIT. We will also determine if the PSEP results in a favorable change in LBP beliefs. The PSEP educates individuals in an evidence-based, psychosocial approach to the management of LBP, which decreases the likelihood of experiencing chronic LBP. We will use a validated self-report questionnaire to measure Soldiers' LBP beliefs regarding outcome and management. We will measure LBP beliefs before and after AIT (a 12-week period).

Study Design: Cluster randomized clinical trial. Twelve companies of Soldiers (n = 2700) reporting to advanced individual training for the 91 W military occupational specialty training will be randomly assigned to CSEP and PSEP (combined education and exercise prevention program), CSEP (exercise prevention program), PSEP and TEP (educational prevention program), and TEP (standard physical training).

Relevance: The results of this study will have several immediate applications for Soldiers. The widespread incorporation of effective preventative strategies will certainly result in a substantial reduction of LBP in the military. Programs that effectively prevent the occurrence and severity of LBP would benefit the U.S. Armed Forces by improving the readiness of their Soldiers, reducing economic burden, and limiting disability among Soldiers. For example, an average cost of $136.02 per LBP visit was calculated for 2004. A 40% reduction in the recurrence of LBP after completing the CSEP would generate a cost savings of $3,343,230 by the 4th fiscal year (approximately 1/5 of the total cost of LBP for one FY).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 35 years old (or emancipated minor)
* Participating in 91 W (combat medic) MOS training
* English speaking and reading

Exclusion Criteria:

* Currently seeking medical care for LBP
* Previous medical history that includes any surgery for LBP (examples include but are not limited to lumbar fusion, lumbar decompression, and lumbar discectomy)
* History of degenerative joint disease, arthritis, spine trauma or vertebral fractures, spondylolisthesis, and congenital spine disorders
* Currently unable to participate in AIT due to injury in foot, ankle, knee, hip, neck, shoulder, elbow, wrist, or hand injury.
* History of fracture (stress or traumatic) in proximal femur and/or pelvis
* Pregnancy (Note: Pregnancy will not result in termination from the study, even though it is an exclusion criteria at enrollment.)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4325 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Episodes of low back pain | 2 years
Duration of low back pain | 2 years
Severity of low back pain | 2 years

SECONDARY OUTCOMES:
Muscle function | 12 weeks
Beliefs about low back pain | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z George, PT, PHD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Brooke Army Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Background] George SZ, Childs JD, Teyhen DS, Wu SS, Wright AC, Dugan JL, Robinson ME. Rationale, design, and protocol for the prevention of low back pain in the military (POLM) trial (NCT00373009). BMC Musculoskelet Disord. 2007 Sep 14;8:92. doi: 10.1186/1471-2474-8-92. PMID 17868436
- [Result] George SZ, Childs JD, Teyhen DS, Wu SS, Wright AC, Dugan JL, Robinson ME. Brief psychosocial education, not core stabilization, reduced incidence of low back pain: results from the Prevention of Low Back Pain in the Military (POLM) cluster randomized trial. BMC Med. 2011 Nov 29;9:128. doi: 10.1186/1741-7015-9-128. PMID 22126534
- [Result] Childs JD, Teyhen DS, Van Wyngaarden JJ, Dougherty BF, Ladislas BJ, Helton GL, Robinson ME, Wu SS, George SZ. Predictors of web-based follow-up response in the Prevention Of Low Back Pain In The Military Trial (POLM). BMC Musculoskelet Disord. 2011 Jun 13;12:132. doi: 10.1186/1471-2474-12-132. PMID 21668961
- [Result] Teyhen DS, George SZ, Dugan JL, Williamson J, Neilson BD, Childs JD. Inter-rater reliability of ultrasound imaging of the trunk musculature among novice raters. J Ultrasound Med. 2011 Mar;30(3):347-56. doi: 10.7863/jum.2011.30.3.347. PMID 21357556
- [Result] Childs JD, Teyhen DS, Casey PR, McCoy-Singh KA, Feldtmann AW, Wright AC, Dugan JL, Wu SS, George SZ. Effects of traditional sit-up training versus core stabilization exercises on short-term musculoskeletal injuries in US Army soldiers: a cluster randomized trial. Phys Ther. 2010 Oct;90(10):1404-12. doi: 10.2522/ptj.20090389. Epub 2010 Jul 22. PMID 20651013
- [Result] Childs JD, Teyhen DS, Benedict TM, Morris JB, Fortenberry AD, McQueen RM, Preston JB, Wright AC, Dugan JL, George SZ. Effects of sit-up training versus core stabilization exercises on sit-up performance. Med Sci Sports Exerc. 2009 Nov;41(11):2072-83. doi: 10.1249/MSS.0b013e3181a84db2. PMID 19812508
- [Result] Robinson ME, Teyhen DS, Wu SS, Dugan JL, Wright AC, Childs JD, Yang G, George SZ. Mental health symptoms in combat medic training: a longitudinal examination. Mil Med. 2009 Jun;174(6):572-7. doi: 10.7205/milmed-d-02-4108. PMID 19585767
- [Result] George SZ, Teyhen DS, Wu SS, Wright AC, Dugan JL, Yang G, Robinson ME, Childs JD. Psychosocial education improves low back pain beliefs: results from a cluster randomized clinical trial (NCT00373009) in a primary prevention setting. Eur Spine J. 2009 Jul;18(7):1050-8. doi: 10.1007/s00586-009-1016-7. Epub 2009 May 6. PMID 19418075
- [Derived] Childs JD, Wu SS, Andrade RL, Bonner VE, Bowman JA, Butler AM, Teyhen DS, George SZ. Incremental Effects of Telephone Call Center and Healthcare Utilization Database Use to Improve Follow-up Rate in the Prevention of Low Back Pain in the Military Trial. US Army Med Dep J. 2015 Oct-Dec:24-30. PMID 26606405
- [Derived] Childs JD, Wu SS, Teyhen DS, Robinson ME, George SZ. Prevention of low back pain in the military cluster randomized trial: effects of brief psychosocial education on total and low back pain-related health care costs. Spine J. 2014 Apr;14(4):571-83. doi: 10.1016/j.spinee.2013.03.019. Epub 2013 Apr 19. PMID 23608562
- See also: Link to abstract and paper for primary study results — http://www.biomedcentral.com/1741-7015/9/128/abstract